CLINICAL TRIAL: NCT03894046
Title: A Randomized, Active-controlled Study to Evaluate the Efficacy and Safety of Intravenous Sulbactam-ETX2514 in the Treatment of Patients With Infections Caused by Acinetobacter Baumannii-calcoaceticus Complex
Brief Title: Study to Evaluate the Efficacy and Safety of Intravenous Sulbactam-ETX2514 in the Treatment of Patients With Infections Caused by Acinetobacter Baumannii-calcoaceticus Complex
Acronym: ATTACK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS2514-2017-0004
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Acinetobacter Baumannii-calcoaceticus Complex; Hospital-acquired Bacterial Pneumonia; Ventilator-associated Bacterial Pneumonia; Bacteremia; Colistin Resistant ABC
MeSH Terms: conditions — Bacteremia | interventions — Sulbactam; durlobactam; Colistin; Imipenem; Cilastatin

STUDY DESIGN:
Masking Description: Study drugs will not be masked due to logistical reasons, every attempt will be made to maintain the blind for patients, all staff at the site, and the Sponsor or its designees, except for the treatment physician and other immediate healthcare providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - Group 1 (Experimental): Part A was the pivotal, assessor-blind, randomized, comparative portion of the study in patients with documented ABC hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), ventilated pneumonia (VP), or bacteremia.
  Part A - Group 1 (experimental): 1.0 g sulbactam/1.0 g durlobactam IV infused over 3 hours every 6 hours (q6h) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h
  Interventions: Drug: Sulbactam; Drug: Durlobactam; Drug: Imipenem/Cilastatin 500 mg/500 mg
- Part A - Group 2 (Active Comparator): Part A - Group 2 (control group): 2.5 mg/kg colistin IV infused over 30 minutes every 12 hours (after an initial loading dose of colistin 2.5 to 5 mg/kg) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h.
  Interventions: Drug: Colistin; Drug: Imipenem/Cilastatin 500 mg/500 mg
- Part B - Group 3 (Experimental): Part B (Group 3) was the open-label, supportive portion of the study that included patients known to have HABP, VABP, VP, and/or bacteremia infections associated with ABC organisms resistant to colistin or polymyxin B, who failed a colistin or polymyxin B regimen prior to study entry or were on acute renal replacement therapy, and patients with infections due to colistin- or polymyxin B-resistant ABC with sources of infection other than HABP, VABP, VP, and/or bacteremia.
  Part B - Group 3: 1.0 g ETX2514/1.0 g sulbactam IV infused over 3 hours q6h plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h.
  Interventions: Drug: Sulbactam; Drug: Durlobactam; Drug: Imipenem/Cilastatin 500 mg/500 mg

INTERVENTIONS:
Drug: Sulbactam — 1.0 g sulbactam IV infused over 3 hours every 6 hours (q6h).
  Arms: Part A - Group 1; Part B - Group 3
Drug: Durlobactam — 1.0 g durlobactam IV infused over 3 hours every 6 hours (q6h).
  Sulbactam-Durlobactam: Treatment for 7 days up to 14 days if clinically indicated.
  Other Names: ETX2514
  Arms: Part A - Group 1; Part B - Group 3
Drug: Colistin — Treatment for 7 days up to 14 days if clinically indicated.
  Other Names: COLOMYCIN INJECTION 2 million IU/vial
  Arms: Part A - Group 2
Drug: Imipenem/Cilastatin 500 mg/500 mg — 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h. Treatment for 7 days up to 14 days if clinically indicated.

SUMMARY:
This is a 2-part study, with Part A being the randomized, controlled portion of the study in patients with ABC hospital-acquired bacterial pneumonia (HABP), ventilator-associated bacterial pneumonia (VABP), or bacteremia. Part B is the single-group portion of the study and includes ABC infections that are resistant to or have failed colistin or polymyxin B treatment, as detailed in the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

PART A

1. A confirmed diagnosis of a serious infection that will require treatment with IV antibiotics;
2. A known infection caused by ABC (bacteremia, HABP, VABP, VP, cUTI or AP, or surgical or post-traumatic wound infections) as either a single pathogen or member of a polymicrobial infection based on evidence from culture or, if available, rapid diagnostic test from a sample collected within 72 hours prior to randomization (HABP/VABP/VP patients), AND 1 of the following:

   1. Has received no more than 48 hrs of potentially effective (ie, Gram negative coverage) antimicrobial therapy prior to the first dose of study drug;
   2. Is clinically failing prior treatment regimens
3. APACHE II score 10 and 30 inclusive, or SOFA score between 7 and 11 inclusive, at time of diagnosis
4. Expectation, in the judgment of the Investigator, that the patient will benefit from effective antibiotic therapy and appropriate supportive care for the anticipated duration of the study
5. Women of childbearing potential (ie, not post-menopausal or surgically sterilized) must have a negative highly sensitive urine or serum pregnancy test before randomization. Participating women of childbearing potential must be willing to consistently use one highly effective method of contraception (ie, condom, combined oral contraceptive, implant, injectable, indwelling intrauterine device, or a vasectomized partner) from Screening until at least 30 days after administration of the last dose of study drug.

PART B

1. Has an infection (HABP, VABP, VP, bacteremia, cUTI, AP, or surgical or post-traumatic wound infections) caused by ABC organisms known to be resistant to colistin (defined as MIC ≥4 mg/L by a non-agar based method);

1. Known to be resistant to colistin or polymyxin B; or
2. Known intolerance to colistin; or
3. Has myasthenia gravis or another neuromuscular syndrome(s) that contraindicates colistin and is not ventilated; or
4. Has acute kidney injury and is receiving renal replacement therapy at study entry.

Exclusion Criteria:

1. Evidence of active concurrent pneumonia requiring additional antimicrobial treatment
2. Presence of suspected or confirmed deep seated bacterial infections such as bacterial Gram negative osteomyelitis, endocarditis, or meningitis requiring prolonged therapy, as determined by history and/or physical examination;
3. Sustained shock with persisting hypotension requiring vasopressors to maintain mean arterial pressure (MAP) ≥ 60 mmHg;
4. Pregnant or breastfeeding women;
5. Receiving peritoneal dialysis;
6. Requirement for continuing treatment with probenecid, methotrexate, ganciclovir, valproic acid, or divalproex sodium during the study;
7. Evidence of significant hepatic disease or dysfunction, including known acute viral hepatitis, hepatic cirrhosis, hepatic failure, chronic ascites, or hepatic encephalopathy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (5):
  - Entasis Research Site, Chicago, Illinois
  - Entasis Research Site, Shreveport, Louisiana
  - Entasis Research Site, Cincinnati, Ohio
  - Entasis Research Site, Memphis, Tennessee
  - Entasis Research Site, Houston, Texas
- Belarus (4):
  - Entasis Research Site, Brest
  - Entasis Research Site, Grodno
  - Entasis Research Site, Homyel
  - Entasis Research Site, Minsk
- Brazil (5):
  - Entasis Research Site, Belo Horizonte
  - Entasis Research Site, Campinas
  - Entasis Research Site, Porto Alegre
  - Entasis Research Site, Salvador
  - Entasis Research Site, São José do Rio Preto
- China (18):
  - Entasis Research Site 1, Beijing
  - Entasis Research Site 2, Beijing
  - Entasis Research Site 3, Beijing
  - Entasis Research Site, Changsha
  - Entasis Research Site, Chongqing
  - Entasis Research Site, Guangzhou
  - Entasis Research Site, Hebei
  - Entasis Research Site 1, Hefei
  - Entasis Research Site 2, Hefei
  - Entasis Research Site, Hubei
  - Entasis Research Site, Nanchang
  - Entasis Research Site, Nanjing
  - Entasis Research Site, Nanning
  - Entasis Research Site 1, Shanghai
  - Entasis Research Site 2, Shanghai
  - Entasis Research Site, Shenzhen
  - Entasis Research Site, Tianjin
  - Entasis Research Site, Wuhan
- Greece (5):
  - Entasis Research Site 1, Athens
  - Entasis Research Site 3, Athens
  - Entasis Research Site, Heraklion
  - Entasis Research Site, Larissa
  - Entasis Research Site, Thessaloniki
- Hungary (3):
  - Entasis Research Site 1, Budapest
  - Entasis Research Site 2, Budapest
  - Entasis Research Site, Debrecen
- India (7):
  - Entasis Research Site, Ahmedabad
  - Entasis Research Site, Belagavi
  - Entasis Research Site 2, Gujrāt
  - Entasis Research Site 1, Gujrāt
  - Entasis Research Site, Hyderabad
  - Entasis Research Site, Kolkata
  - Entasis Research Site, Pune
- Israel (4):
  - Entasis Research Site, Holon
  - Entasis Research Site, Tel Aviv
  - Entasis Research Site, Tel Litwinsky
  - Entasis Research Site, Ẕerifin
- Lithuania (3):
  - Entasis Research Site, Kaunas
  - Entasis Research Site, Klaipėda
  - Entasis Research Site, Vilnius
- Mexico (5):
  - Entasis Research Site 1, Guadalajara
  - Entasis Research Site 2, Guadalajara
  - Entasis Research Site, Mexico City
  - Entasis Research Site, Monterrey
  - Entasis Research Site, San Luis Potosí City
- Peru (5):
  - Entasis Research Site, Bellavista
  - Entasis Research Site, Cusco
  - Entasis Research Site, Lima
  - Entasis Research Site, San Isidro
  - Entasis Research Site, San Martín de Porres
- Entasis Research Site, Ponce, Puerto Rico
- Russia (9):
  - Entasis Research Site, Arkhangelsk
  - Entasis Research Site, Krasnodar
  - Entasis Research Site 1, Novosibirsk
  - Entasis Research Site 2, Novosibirsk
  - Entasis Research Site 3, Novosibirsk
  - Entasis Research Site 2, Saint Petersburg
  - Entasis Research Site, Smolensk
  - Entasis Research Site 1, Tomsk
  - Entasis Research Site 2, Tomsk
- South Korea (3):
  - Entasis Research Site, Gyeonggi-do
  - Entasis Research Site 1, Seoul
  - Entasis Research Site 2, Seoul
- Taiwan (3):
  - Entasis Research Site, Kaohsiung City
  - Entasis Research Site, Taichung
  - Entasis Research Site, Taipei
- Thailand (4):
  - Entasis Research Site, Chiang Mai
  - Entasis Research Site, Khon Kaen
  - Entasis Research Site, Nakhon Ratchasima
  - Entasis Research Site, Nonthaburi
- Turkey (Türkiye) (6):
  - Entasis Research Site 1, Ankara
  - Entasis Research Site 2, Ankara
  - Entasis Research Site, Eskişehir
  - Entasis Research Site, Kocaeli
  - Entasis Research Site, Küçükçekmece
  - Entasis Research Site, Trabzon

REFERENCES:
- [Derived] Kaye KS, Shorr AF, Wunderink RG, Du B, Poirier GE, Rana K, Miller A, Lewis D, O'Donnell J, Chen L, Reinhart H, Srinivasan S, Isaacs R, Altarac D. Efficacy and safety of sulbactam-durlobactam versus colistin for the treatment of patients with serious infections caused by Acinetobacter baumannii-calcoaceticus complex: a multicentre, randomised, active-controlled, phase 3, non-inferiority clinical trial (ATTACK). Lancet Infect Dis. 2023 Sep;23(9):1072-1084. doi: 10.1016/S1473-3099(23)00184-6. Epub 2023 May 11. PMID 37182534

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The total number of participants enrolled in the study was 207. However, two (2) patients were transferred from Part A to part B. These participants were analyzed at each arm until/ from the time point of transfer.
Groups:
- Part A - Group 1: Experimental.
  1.0 g sulbactam/1.0 g durlobactam IV infused over 3 hours every 6 hours (q6h) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h;
- Part A - Group 2: Control group.
  2.5 mg/kg colistin IV infused over 30 minutes every 12 hours (after an initial loading dose of colistin 2.5 to 5 mg/kg) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h.
- Part B - Group 3: Experimental.
  Group 3: 1.0 g ETX2514/1.0 g sulbactam IV infused over 3 hours q6h plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h.
Period: Overall Study
Arm/Group | Part A - Group 1 | Part A - Group 2 | Part B - Group 3
Started | 92 | 89 | 26
Completed | 69 | 61 | 20
Not Completed | 23 | 28 | 6
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Death | 15 | 21 | 4
Not completed — No growth of ABC | 2 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Prohibited concomitant medication | 1 | 0 | 0
Not completed — Transferred to other arm/group | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Two (2) participants were transferred from Part A to part B. These participants were analyzed at each arm until/ from the time point of transfer. The number of participants is reported according to the initial Arm/group in which individual participant was assigned.
Groups:
- Part A- Group 1: Experimental. Group 1 (experimental): 1.0 g sulbactam/1.0 g durlobactam IV infused over 3 hours every 6 hours (q6h) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h;
- Part A - Group 2: Control Group (active comparator). Group 2 (control group): 2.5 mg/kg colistin IV infused over 30 minutes every 12 hours (after an initial loading dose of colistin 2.5 to 5 mg/kg) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h.
- Total: Total of all reporting groups
Arm/Group | Part A- Group 1 | Part A - Group 2 | Part B - Group 3 | Total
Number analyzed (Participants) | 92 | 89 | 26 | 207
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 37 | 18 | 98
  >=65 years | 49 | 52 | 8 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (15.42) | 66.9 (17.13) | 56.2 (16.33) | 59.8 (16.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 5 | 52
  Male | 68 | 66 | 21 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 0 | 7
  Asian | 33 | 44 | 3 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 48 | 41 | 23 | 112
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With All-Cause Mortality in CRABC m-MITT Population
Description: The primary efficacy endpoint for the study is 28-day all-cause mortality in the CRABC m-MITT population in Part A.
Time Frame: 28 Days
Population: CRABC m-MITT (Carbapenem-resistant Acinetobacter baumannii-calcoaceticus complex Microbiologically Modified Intent-to-Treat Population).
  The CRABC m-MITT Population included patients who met m-MITT criteria and had a baseline ABC organism that was confirmed to be carbapenem-resistant (MIC of imipenem/meropenem ≥8 ug/mL) by the central laboratory or by the local laboratory.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - Group 1: Experimental.
  Group 1 (experimental): 1.0 g sulbactam/1.0 g durlobactam IV infused over 3 hours every 6 hours (q6h) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h;
Arm/Group | Part A - Group 1 | Part A - Group 2
Number analyzed (Participants) | 63 | 62
Participants | 12 | 20
Statistical Analysis 1: Comparison: Part A - Group 1 vs Part A - Group 2; The non-inferiority assessment was based on the 2-sided 95% CIs computed using a continuity-corrected Z-statistic for the difference ([sulbactam-durlobactam + imipenem/cilastatin] - [colistin + imipenem/cilastatin]) in 28-day all-cause mortality rates between the treatment groups; Test type: Non-Inferiority — Non-inferiority was concluded if the upper limit of the 2-sided 95% CI was less than +20%. Superiority was concluded if the upper limit of the 2-sided 95% CI was less than 0; Mean Difference (Final Values) = -13.2, 95% CI 2-sided [-30 to 3.5]

2. Primary Outcome: Proportion of Patients With Nephrotoxicity
Description: The primary safety endpoint for the study is nephrotoxicity, as measured by the Risk-Injury-Failure-Loss-End-stage renal disease (RIFLE) criteria, in the MITT population in Part A.
Time Frame: 28 days
Population: MITT (Modified Intent To Treat population containing all patients who received any amount of study drug).
  Analysis of patients with nephrotoxicity as measured by RIFLE criteria at any post-baseline visit based on the Investigator's opinion for the Safety Population for Part A, excluding patients with chronic hemodialysis at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - Group 1 | Part A - Group 2
Number analyzed (Participants) | 91 | 85
Participants | 12 | 32
Statistical Analysis 1: Comparison: Part A - Group 1 vs Part A - Group 2; Analysis of patients with nephrotoxicity as measured by RIFLE criteria at any post-baseline visit based on the Investigator's opinion for the Safety Population for Part A, excluding patients with chronic hemodialysis at baseline baseline; Test type: Other; p = 0.0002, Chi-squared — p-value was obtained based on a Chi-Square test for treatment group differences

ADVERSE EVENTS:
Time Frame: Adverse event monitoring starts from the time the patient consents to the study until up to 30 days after treatment.
Description: A Treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that occurred on or after the administration of the first dose of study drug.
  NOTE: Total Number of Participants at Risk includes participants who received at least one dose of the study treatment. This also applies to Serious and Other (Not Including Serious) Adverse Events described below.
Groups:
- Part A - Group 1: Experimental. Group 1 (experimental): 1.0 g sulbactam/1.0 g durlobactam IV infused over 3 hours every 6 hours (q6h) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h;
  In total, 91 patients received any amount of study drug treatment in Part A - Group 1 and were considered the Safety Population for this group.
- Part A - Group 2: Control group (active comparator). Group 2 (control group): 2.5 mg/kg colistin IV infused over 30 minutes every 12 hours (after an initial loading dose of colistin 2.5 to 5 mg/kg) plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h.
  In total, 86 patients received any amount of study drug treatment in Part A - Group 2 - control group and were considered the Safety Population for this group.
- Part B - Group 3: Experimental. Group 3: 1.0 g ETX2514/1.0 g sulbactam IV infused over 3 hours q6h plus 1.0 g imipenem/1.0 g cilastatin IV infused over 1 hour q6h.
  There were 28 patients who received any amount of study drug in Part B and were included in the Safety Population for Part B.
Arm/Group | Part A - Group 1 | Part A - Group 2 | Part B - Group 3
All-Cause Mortality (participants affected / at risk) | 25/91 | 31/86 | 4/28
Serious Adverse Events (participants affected / at risk) | 36/91 | 42/86 | 9/28
Other Adverse Events (participants affected / at risk) | 48/91 | 53/86 | 14/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Group 1 (N=91) | Part A - Group 2 (N=86) | Part B - Group 3 (N=28)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 4 (4) | 2 (2)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Weaning failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 4 (4) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Primary biliary cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 7 (9) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Acinetobacter infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - Group 1 (N=91) | Part A - Group 2 (N=86) | Part B - Group 3 (N=28)
Hypotension (Vascular disorders) | 5 (5) | 5 (5) | 1 (1)
Pyrexia (General disorders) | 9 (14) | 8 (11) | 1 (1)
Blood creatinine increased (Investigations) | 2 (6) | 7 (10) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Enterococcus test positive (Investigations) | 0 (0) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 12 (18) | 11 (13) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 15 (16) | 9 (11) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (7) | 5 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 9 (12) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (21) | 9 (19) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (11) | 8 (9) | 1 (1)
Tracheobronchitis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (2) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 6 (9) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03894046/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03894046/SAP_001.pdf